CLINICAL TRIAL: NCT02827812
Title: Home-Based Telesurveillance and Rehabilitation Program in Parkinson's Disease: Pilot Randomized Trial
Brief Title: Telemedicine Program in Parkinson's Disease (TELEPARK)
Acronym: TELEPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Fabrizio Pisano, Head of Neurological Rehabilitation Division, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1_neuro_veruno
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants Telemedicine Care (PTE) (Experimental): A. Comprehensive evaluation at baseline (T0) and at the end of the study (T1).
  B. Physical Intervention at home for 60 minutes 3 days/week for three months
  C. Home-Based telemedicine program:
  Interventions: Other: Comprehensive evaluation; Other: Physical Intervention at home; Other: Home-Based telemedicine program
- Participants Usual Care (PUC) (Active Comparator): A. Comprehensive evaluation at baseline (T0) and at the end of the study (T1).
  B. Physical Intervention at home for 60 minutes 3 days/week for three months
  Interventions: Other: Comprehensive evaluation; Other: Physical Intervention at home

INTERVENTIONS:
Other: Comprehensive evaluation — At baseline (T0) and after 3-months (T1) all patients will be evaluated with Scales and questionnaire.
Other: Physical Intervention at home — A traditional custom-tailored rehabilitative exercise program. The exercises will include functional strengthening, stretching, postural changes and balance activities; - An aerobic training on a cycle ergometer 3 days /week for three months.
Other: Home-Based telemedicine program — 1. A nurse-tutor will follow patients through structured telephone appointments, collecting information about disease status and symptoms, offering advice regarding diet, lifestyle and medications and suggesting changes in therapy, according with the neurologist. The patient's clinical data and any suggestions made will be filled in a personal health electronic record.
  2. A physiotherapist-tutor will supervise the patient's home-based individualized rehabilitation program, through scheduled videoconferences.
  Arms: Participants Telemedicine Care (PTE)

SUMMARY:
Parkinson's disease (PD) is a chronic neurodegenerative disease due to the loss of dopaminergic neurons in the substantia nigra, leading to motor symptoms of tremor, rigidity, and bradykinesia, as well as an array of non-motor symptoms that affect cognition, sleep, behaviour, and the autonomic nervous system.

Lifelong rehabilitation measures, along with medication treatment, are the major components of patient management. Physical exercises positively affect patients' quality of life (QOL) and their functional capacities. Poor adherence to rehabilitation, limited patient education, and access to specialized care can be barriers to treatment. A number of papers in fact report that telemedicine is an acceptable means of care delivery reduces travel burdens and may improve patient outcomes. However, most of these studies were not randomized or controlled and did not include nursing home patients, who may benefit the most from specialty care.

Moreover, there is no evidence supporting the use of telerehabilitation for physical assessments of people with PD. For this reason investigators hypothesize that a home telerehabilitation system guiding patients in following their exercise program combined with a computerized decision-support tool monitoring patient performance, would be feasible for and acceptable to patients with PD and would improve functional status.

DETAILED DESCRIPTION:
Aim of the study:

1. Demonstrate the feasibility of at home telesurveillance and rehabilitation program
2. Demonstrate the effectiveness of the program in improving quality of life and functional aspects in patients affected by Parkinson's disease

30 patients affected by Parkinson's disease (PD), will be consecutively screened. The method of sequence generation relied on a computerized random number generator. The person who allocated patients to the two groups was not involved either in treatment or in evaluation of the patients.

The study was submitted for approval of the Central Ethics Review Board. Participants will be randomly assigned to two different groups of training using a random number table to receive either telemedicine care (PTE) or their usual care (PUC).

All the patients will receive in our Institute a comprehensive baseline evaluation conducted by both the neurologist and the physical therapist specialized in the treatment of PD.

During the baseline evaluation (T0), both PTE and PUC will perform two supervised familiarization sessions using the same training protocol to be used once at home.

Caregivers are an essential part in the PD patients' home management and rehabilitation and they therefore will be involved in all educational stages.

Each patient of both groups will receive two types of physical intervention:

1. A traditional custom-tailored rehabilitative exercise program; he will be trained by the therapist on how to perform the exercises. These exercises will include functional strengthening, stretching, postural changes and balance activities
2. An aerobic training All patients will be asked to perform these exercises for 60 minutes 3 days/week for three months.

The training phase will last 20 minutes during the first month and 30 minutes over the second and third month; Training intensity could be progressively increased over the three months of intervention, Aerobic training familiarization sessions will be performed on the same ergometer they will receive for home-based training.

ELIGIBILITY:
Inclusion Criteria:

* 30 patients affected by Parkinson's disease (PD), according to the United Kingdom Parkinson's Disease Society Brain Bank Criteria (Hughes et al.,1992), will be consecutively screened. Participants should have a Hoehn & Yahr stage between 1,5 and 3. All subjects will be on stabilized treatment with L-dopa or dopamine agonists.

All participants will provide written informed consent to the study.

Exclusion Criteria:

* inability to participate in the exercise programs, other neurological conditions in addition to PD, psychiatric complications or personality disorders, musculoskeletal or cardiopulmonary conditions affecting mobility, and non-consent to participate in the study A cognitive impairment scores measured with Mini Mental State Examination (MMSE) ≤ 26/30.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants in the PTE group who will concluded the home-based program. | Through study completion, an average of 3 months
  The program is feasible if at least 80% of participants in the PTE group complete the home program lasting 3 months. The participant completes the home program if carries out at least 50% of the prescribed physical activity.

SECONDARY OUTCOMES:
Improvement of quality of life (QoL) measured by the "Parkinson's disease questionnaire" (PDQ-39) | Difference between two groups of PDQ-39 measured at baseline (T0) and after 3 months (T1)
  The PDQ consider eight discrete scales on mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communication (3 items) and bodily discomfort (3 items). Participants are asked to indicate the frequency of each event by selecting one of 5 options (from never to always). Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL
Improvement of exercise tolerance capacity measured in the meters walked, by the 6-min walk test (6MWT) | Difference between two groups of 6MWT measured at baseline (T0) and after 3 months (T1)
Improvement of balance measured by Balance Evaluation Systems Test (Mini BesTest) | Difference between two groups of Mini BesTest measured at baseline (T0) and after 3 months (T1)
  The Mini-BESTest includes 14 items representing four domains of dynamic balance:anticipatory postural adjustments (items 1-3), postural responses (items 4-6), sensory orientation (items 7-9) and balance during gait (items 10-14). The Mini-BESTest items are rated on a 3-point scale from 0 to 2 and the total score ranges from 0 to 28 with a higher score indicating better balance performance.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schwab S, Vatankhah B, Kukla C, Hauchwitz M, Bogdahn U, Furst A, Audebert HJ, Horn M; TEMPiS Group. Long-term outcome after thrombolysis in telemedical stroke care. Neurology. 2007 Aug 28;69(9):898-903. doi: 10.1212/01.wnl.0000269671.08423.14. PMID 17724293
- [Result] Scalvini S, Zanelli E, Comini L, Dalla Tomba M, Troise G, Febo O, Giordano A. Home-based versus in-hospital cardiac rehabilitation after cardiac surgery: a nonrandomized controlled study. Phys Ther. 2013 Aug;93(8):1073-83. doi: 10.2522/ptj.20120212. Epub 2013 Apr 18. PMID 23599353
- [Result] Hubble JP, Pahwa R, Michalek DK, Thomas C, Koller WC. Interactive video conferencing: a means of providing interim care to Parkinson's disease patients. Mov Disord. 1993 Jul;8(3):380-2. doi: 10.1002/mds.870080326. PMID 8341308
- [Result] Samii A, Ryan-Dykes P, Tsukuda RA, Zink C, Franks R, Nichol WP. Telemedicine for delivery of health care in Parkinson's disease. J Telemed Telecare. 2006;12(1):16-8. doi: 10.1258/135763306775321371. PMID 16438773
- [Result] Biglan KM, Voss TS, Deuel LM, Miller D, Eason S, Fagnano M, George BP, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Dorsey ER. Telemedicine for the care of nursing home residents with Parkinson's disease. Mov Disord. 2009 May 15;24(7):1073-6. doi: 10.1002/mds.22498. PMID 19353687
- [Result] Arcolin I, Pisano F, Delconte C, Godi M, Schieppati M, Mezzani A, Picco D, Grasso M, Nardone A. Intensive cycle ergometer training improves gait speed and endurance in patients with Parkinson's disease: A comparison with treadmill training. Restor Neurol Neurosci. 2016;34(1):125-38. doi: 10.3233/RNN-150506. PMID 26684265